CLINICAL TRIAL: NCT00265044
Title: Innovations to Implementing Evidence-based Clinical Practice
Brief Title: Improving Practice Patterns for the Treatment of Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: IMV 04-091
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2006-05

CONDITIONS: Hypertension
Keywords: Behavior Change; patient Education
MeSH Terms: conditions — Hypertension | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Provider Education; Behavioral: Hypertension Alert; Behavioral: Patient Education

INTERVENTIONS:
Behavioral: Provider Education
Behavioral: Hypertension Alert
Behavioral: Patient Education

SUMMARY:
To improve the quality of hypertension care in our facility, while concurrently, examining the relative contribution of each aspect of a multi-factorial intervention designed to improve hypertension care.

DETAILED DESCRIPTION:
This project was a randomized trial designed to examine the relative contribution of three quality improvement interventions of increasing intensity on BP control in veterans. Providers in each stratum and their eligible patients were randomized to one of three study arms. The providers randomized to the first arm received education alone, and were considered the controls. Providers randomized to the second arm received both provider education and a hypertension alert. The third arm included provider education, a hypertension alert, and patient education. Patients were eligible for inclusion if they were aged 21- 90 years and filled their medications with the VA pharmacies. Between July and December 2003, we determined patient eligibility using a search strategy using data from the Mid South Quality Improvement Data warehouse, which is downloaded monthly from Veterans' Health Information System and Technology Architecture (VistA).

ELIGIBILITY:
Inclusion Criteria:

Patients were eligible for inclusion if they were aged 21- 90 years and filled their medications with the VA pharmacies. Seen in 2003 and had a primary care visit coded as hypertension using International Classification of Diseases Ninth Revision; Clinical Modification (ICD 9-CM) (24) of 401.1 or 401.9 and who were prescribed only one antihypertensive medication

Exclusion Criteria:

More than one antihypertensive medication Refuse consent to review medical record Pregnant Prisoners

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2004-01; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Reaching Systolic BP goal 6 months after intervention

SECONDARY OUTCOMES:
Reaching Diastolic BP goal 6 months after intervention Any additional prescriptions of antihypertensive medications.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Speroff, PhD, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN; Christianne L Roumie, BA MD MPH, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN; Vincent Alvarez, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (1):
- Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee, United States

REFERENCES:
- [Result] Roumie CL, Elasy TA, Greevy R, Griffin MR, Liu X, Stone WJ, Wallston KA, Dittus RS, Alvarez V, Cobb J, Speroff T. Patient education adds critical boost to hypertension management. [Editorial]. VA Research Currents. 2006 Sep 1; 7-8.
- [Result] Roumie CL, Elasy TA, Greevy R, Griffin MR, Liu X, Stone WJ, Wallston KA, Dittus RS, Alvarez V, Cobb J, Speroff T. Improving blood pressure control through provider education, provider alerts, and patient education: a cluster randomized trial. Ann Intern Med. 2006 Aug 1;145(3):165-75. doi: 10.7326/0003-4819-145-3-200608010-00004. PMID 16880458